CLINICAL TRIAL: NCT02050126
Title: Caesarean Scar Revision With the UltraPulse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lumenis Be Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LUM-ABU-UP-12-02
Record Dates: First submitted 2014-01-28; First posted 2014-01-30 (Estimated); Last update posted 2016-04-22 (Estimated); Status verified 2016-04

CONDITIONS: Scar Revision

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Scar Revision (Experimental): Caesarean Scar Revision using Lumenis UltraPulse Encore.
  Interventions: Device: Lumenis UltraPulse Encore.

INTERVENTIONS:
Device: Lumenis UltraPulse Encore. — Treatment using Lumenis UltraPulse Encore.

SUMMARY:
Ten (10) adult female subjects that had a caesarean surgery performed.Study will be conducted in 1 site.

Each subject will receive three treatments on one area that was randomly chosen. The other area will be left untreated and will serve as a control.

The objective is to Evaluate the clinical impact of UltraPulse fractional carbon dioxide laser treatment on the appearance of a Caesarean Scar (CS) as compared to a similar untreated scar side.

ELIGIBILITY:
Inclusion Criteria:

1. Females in good general health older than 22 years of age and younger than 55 years of age.
2. Presenting with a caesarean scar mature and stable caesarean scar (at least 1 year post procedure).
3. At least six months following termination of breast feeding.
4. Willing to give and sign an informed consent form and a photographic release form.
5. Willing to comply with study dosing and complete the entire course of the study .
6. Performed negative pregnancy test.

Exclusion Criteria:

1. Active bacterial, fungal, or viral infection in the treatment area.
2. Active cold sores, or herpes in the treatment area.
3. Recent excessive exposure to sunlight or artificial UV light (e.g.: use of tanning beds/booths and/or sunbathing) or expectations of tanning during the time of the study .
4. History of or the presence of any skin condition/disease that might interfere with the diagnosis or evaluation of study parameters (i.e., atopic dermatitis, eczema, psoriasis).
5. Treatment with a systemic retinoid within the past year (e.g., Accutane®, Roche Dermatologics).
6. History or presenting with a keloid scar.
7. Any current or recent treatment for cancer.
8. Any uncontrolled systemic disease. A potential subject in whom therapy for a systemic disease is not yet stabilized will not be considered for entry into the study.
9. Significant history or current evidence of a medical, psychological or other disorder that, in the investigator's opinion, would preclude enrollment into the study.
10. Previous laser treatments on the same scar at least 0.5 year prior to this evaluation.
11. Subject planning any other cosmetic procedure to the study area during the study period, other than the treatments that will be performed by the investigator .
12. Any other condition that may exclude patient for treatment per physician discretion.
13. Female subject who is pregnant, nursing an infant .

Ages: 22 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2013-04; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Scar Evaluation | 3 month following the 3rd treatment.
  VSS , POSAS, Appearance assessment-Evaluation of the scar by blinded investigator.

SECONDARY OUTCOMES:
Scar Evaluation. | At base line , at the 3rd treatment and at the 1, 3 and 6 months follow-up
  VSS assessment -Evaluation of the scar by blinded investigator.
POSAS assessment | At base line , at the 3rd treatment and at the 1, 3 and 6 months follow-up
  POSAS assessment by blinded Investigator and subject
Scar Thickness and Uniformity | At base line, at the 3rd treatment and at the 1, 3 and 6 months follow-up
  A High Definition Ultrasound (US) device will be used to generate a high resolution image of the skin layers of the treated and non-treated scar in order to measure and compare changes in scar thickness and uniformity.
Scar color | At base line, at the 3rd treatment and at the 1, 3 and 6 months follow-up.
  Colorimeter will be used for color measurement.
Histochemical Changes in scar tissue | Immediately before the 2nd, and 3rd treatment
  Histochemical analysis of scar tissue with different staining for analysis of changes following treatment:
  * H&E staining and histology for collagen arrangement, epidermal rete ridges and measurement of scar depth
  * Collagen type I and III staining
  * Elastin staining
  * Immunohistochemistry for TGF-beta 1, 2, 3 and MMPs
Subject's satisfaction | At the 3rd treatment and at the 1, 3 and 6 month follow-up
  Subject's satisfaction of the treatment using a Satisfaction Scale as follows: None; Slight; Moderate; Good; Very Good.

CONTACTS AND LOCATIONS:
Overall Officials: Merete Hædersdal, dr. med., ph.d., Principal Investigator — Dermato-venerologisk Afdeling D42
Locations (1):
- Dermato-venerologisk Afdeling D42, Copenhagen, Bispebjerg Bakke 23, Denmark